CLINICAL TRIAL: NCT02971085
Title: Seoul National University Prospectively Enrolled Registry for Prostate Cancer With Active Surveillance
Acronym: SUPER-PC-AS
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chang Wook Jeong, Professor, Seoul National University Hospital
Other Study IDs: 2016-2957
Record Dates: First submitted 2016-11-13; First posted 2016-11-22 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
Keywords: low-risk prostate cancer; active surveillance; pathologic reclassification
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Active surveillance: This is the prospective cohort study with single group of active surveillance. We define our cohort group as the patients with following criteria: Men < 80 years, pathologically proven adenocarcinoma of the prostate by transrectal prostate biopsy ≥ 10 cores, pre-biopsy PSA ≤ 10ng/ml, PSA density < 0.15 ng/ml/ml, clinical stage T1-2a, biopsy Gleason score ≤ 6, number of positive cores ≤ 2, maximum cancer involvement in any one core ≤ 20%, and no PIRADS 5 lesion on multiparametric prostate MRI (1.5T or 3T).
  Interventions: Procedure: Active surveillance

INTERVENTIONS:
Procedure: Active surveillance — Active surveillance cohorts are routinely performed the systematic biopsy ≥ 12 cores by TRUS-guided or MR-TRUS fusion according to the protocol based by time path as 1, 2, 4, 7, 10 years and subsequently every 5 years following initial TRUS biopsy.

SUMMARY:
In this study, the investigators aim to establish the prostate cancer active surveillance prospective cohort in our institution, and finally investigate the 5 year rates of reclassification during active surveillance as the primary endpoint of the current study.

DETAILED DESCRIPTION:
Prostate cancer (PCa) remains one of the most commonly diagnosed malignancies in men worldwide. Early diagnosis and definitive therapy seem to improve oncological outcomes in men with high-risk disease, but significant concerns exist in terms of the overdiagnosis and overtreatment of patients with lower-risk tumors. In this context, active surveillance (AS) has recently emerged as a alternative treatment strategy in PCa patients with low risk cancers. However, published data are based on Western population with different protocol, and therefore; well-controlled data with well-organized and prospective cohort are urgently needed in Korean patients with low-risk PCa because Korean patients have significantly different tumor characteristics compared to Western patients. Here, the investigators have a plan to establish the Seoul National University Enrolled Registry for Prostate Cancer with Active Surveillance, and finally provide the concrete evidence for the clinical outcomes of active surveillance program as the primary therapeutic strategy for low-risk PCa in Korean men.

ELIGIBILITY:
Inclusion Criteria:

1. Men < 80 years
2. Pathologically proven adenocarcinoma of the prostate by transrectal prostate biopsy ≥ 10 cores
3. Pre-Bx PSA ≤ 10ng/ml
4. PSA density < 0.15ng/ml/ml
5. Clinical stage T1-2a
6. Biopsy Gleason score ≤ 6
7. No. of positive cores ≤ 2
8. Maximum cancer involvement in any one core ≤ 20%.
9. No PIRADS 5 lesion on multiparametric prostate MRI (1.5T or 3T)
10. Participants must be willing to attend the follow-up visits - T1a-b disease should be confirmed by systematic TRUS-Bx ≥ 10 cores

Exclusion Criteria:

1. A former therapy for prostate cancer.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean men with pathologically proven adenocarcinoma of prostate cancer with low-risk who will be treated by active surveillance protocol in Seoul National University Hospital.
Sampling Method: Probability Sample
Enrollment: 410 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Pathological reclassification | 5 year
  5-year rate of pathological reclassification during active surveillance

SECONDARY OUTCOMES:
active treatment-free survival | 1, 3, 5, 7, 10 years
  active treatment-free survival rate
metastasis-free survival | 3, 5, 10 years
  metastasis-free survival rate
overall survival | 3, 5, 10 years
  overall survival rate
rates of active surveillance maintenance | 1, 3, 5, 7, 10 years
  rates of active surveillance maintenance
HRQoL scores (measured by EPIC-CP) | 1, 3, 5, 7, 10 years
  HRQoL scores (measured by EPIC-CP)
Utility value (measured by EQ-5D-5L) | 1, 3, 5, 7, 10 years
  Utility value (measured by EQ-5D-5L)

CONTACTS AND LOCATIONS:
Overall Officials: Chang Wook Jeong, M.D, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided